CLINICAL TRIAL: NCT01942525
Title: Intrauterine Growth Restriction Has an Impact on Amplitude-integrated EEG in Preterm Infants
Brief Title: Influence of Intrauterine Growth Restriction on Amplitude-integrated EEG in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Katrin Klebermass-Schrehof, MD, Medical University of Vienna
Other Study IDs: KKS-07-2013
Record Dates: First submitted 2013-08-24; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Intrauterine Growth Restriction; Premature - Weight 1000g-2499g or Gestation of 28-37weeks; Neurodevelopmental Disorder; EEG; Spikes, Centrotemporal, Epilepsy of Childhood
Keywords: IUGR; aEEG; preterm infants; neurodevelopmental outcome
MeSH Terms: conditions — Fetal Growth Retardation; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intrauterine growth restriction: birth weight <10th percentile first intervention: aEEG second intervention: assessment of neurodevelopmental follow-up
  Interventions: Other: aEEG
- Appropriate for gestation age: control group with birth weight >10th percentile first intervention: aEEG second intervention: assessment of neurodevelopmental follow-up
  Interventions: Other: aEEG

INTERVENTIONS:
Other: aEEG — The amplitude integrated EEG was performed using a single-channel, biparietal aEEG (CFM 6000; Natus Medical Incorporated, San Carlos, CA)
  Other Names: assessment of neurodevelopmental follow-up

SUMMARY:
Objective: The impact of intrauterine growth restriction (IUGR) on perinatal morbidity and long-term neurodevelopmental outcome has been published in numerous studies. Throughout this analysis, the influence of IUGR on the postnatal amplitude-integrated EEG (aEEG) in preterm infants below 30 weeks of gestation was assessed. The second concern was the correlation between the pattern of the aEEG in the first two weeks with neurodevelopmental outcome, comparing infants with and without IUGR.

Methods: Routinely assessed aEEG data of preterm infants with IUGR born below 30 weeks of gestation in the years 2005 until 2007 were analysed retrospectively according to the aEEG score (combining occurrence of sleep-wake-cycles, background activity and suspected seizure activity). Neurodevelopmental outcome was evaluated at 24 months using the Bayley Scales of Infant Development and standardized neurologic examination.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants below 30 weeks of gestation

Exclusion Criteria:

* congenital anomalies
* severe asphyxia

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Retrospectively, children with intrauterine growth restriction (defined as a birth weight below the 10th percentile) treated at the Neonatal Intensive Care Unit (NICU) of the Medical University Vienna between 2005 and 2007 were included in the study. Besides IUGR, inclusion criteria were gestational age between 23+1 and 29+6 weeks and routinely assessed aEEG measurements. Infants with congenital anomalies and severe asphyxia were excluded. The control group consists of infants of the same age with normal birth weight (>10th percentile) in the same study period.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
aEEG score (including background pattern, occurrence of sleep-wake-cycling and presence of seizure activity) | first 14 days of life
  composite score background activity (BA), occurrence of sleep-wake-cycling (SWC) and presence of seizure activity (SA) meaning score 1= normal (normal BA, SWC yes, SA no) and score 2 and 3 = abnormal (2=abnormality in 1 category (BA, SWC or SA) and score 3= abnormality in 2 or 3 categories

SECONDARY OUTCOMES:
Neurodevelopmental outcome | 24 months
  composite score: Bayley Scales of Infant Development (>85= normal, <70 severely impaired, 71-84= mildly impaired) and standardized neurologic examination (normal or abnormal)

OTHER OUTCOMES:
Morbidity, mortality and neurodevelopmental outcome of patients with IUGR compared to controls | 24 months
  morbidities until discharge (Intraventricular hemorrhage, retinopathy, chronic lung disease, necrotizing enterocolitis, periventricular leucomalacia); mortality and neurodevelopmental outcome (via Bayley Scales of Infant Development >85= normal, <70 = severly impaired)

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Klebermass-Schrehof, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria